CLINICAL TRIAL: NCT01708590
Title: A Phase 3 Study to Evaluate the Efficacy, Safety, and Effect of Withdrawal and Retreatment With Brodalumab in Subjects With Moderate to Severe Plaque Psoriasis: AMAGINE-1
Brief Title: Efficacy, Safety, and Withdrawal and Retreatment With Brodalumab in Moderate to Severe Plaque Psoriasis Subjects
Acronym: AMAGINE-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120102; 2012-000651-13 (EudraCT Number)
Record Dates: First submitted 2012-09-10; First posted 2012-10-17 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Psoriasis
Keywords: psoriasis, brodalumab (AMG 827)
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 210 mg brodalumab (Experimental): Administered by subcutaneous (SC) injection until week 12. At week 12, participants are rerandomized to placebo or continued treatment. Participants are retreated at return of disease.
  Interventions: Drug: 210 mg brodalumab; Drug: placebo
- 140 mg brodalumab (Experimental): Administered by subcutaneous (SC) injection until week 12. At week 12, participants are rerandomized to placebo or continued treatment. Participants are retreated at return of disease.
  Interventions: Drug: 140 mg brodalumab; Drug: placebo
- placebo (Placebo Comparator): Administered by SC injection until week 12. At week 12 particpants are assigned to 210 mg brodalumab.
  Interventions: Drug: 210 mg brodalumab; Drug: placebo

INTERVENTIONS:
Drug: 210 mg brodalumab — 210 mg brodalumab administered subcutaneous (SC)
  Other Names: Siliq
  Arms: 210 mg brodalumab; placebo
Drug: 140 mg brodalumab — 140 mg brodalumab administered subcutaneous (SC)
  Other Names: Siliq
  Arms: 140 mg brodalumab
Drug: placebo — Placebo administered subcutaneous (SC)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of brodalumab taken every two weeks at two different doses.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety and efficacy of brodalumab taken every two weeks at two different doses in participants with moderate to severe plaque psoriasis. A second purpose of this study is to assess the safety and efficacy when brodalumab is replaced with placebo in some participants compared with the participants who are still receiving the brodalumab.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had stable moderate to severe plaque psoriasis for at least 6 months
* Subject must be considered, in the opinion of the investigator, to be a suitable candidate for treatment with a biologic per regional labeling
* Subject has involved body surface area (BSA) ≥ 10%, PASI ≥ 12, and sPGA ≥ 3 at screening and at baseline

Exclusion Criteria:

* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, or other skin conditions at (eg, eczema) that would interfere with study evaluations
* Subject has known history of Crohn's disease
* Subject has any other significant concurrent medical condition or laboratory abnormalities, as defined in the study protocol
* Subject has stopped using certain psoriasis therapies as defined in the study protocol
* Subject has previously used any anti-IL-17 biologic therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (71):
- United States (31):
  - Research Site, Phoenix, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Encino, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, San Ramon, California
  - Research Site, Santa Monica, California
  - Research Site, Alpharetta, Georgia
  - Research Site, West Dundee, Illinois
  - Research Site, Richmond, Kentucky
  - Research Site, Columbia, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fort Gratiot, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Buffalo, New York
  - Research Site, Forest Hills, New York
  - Research Site, Rochester, New York
  - Research Site, Stony Brook, New York
  - Research Site, Wilmington, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Rapid City, South Dakota
  - Research Site, Goodlettsville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
- Canada (10):
  - Research Site, Surrey, British Columbia
  - Research Site, Moncton, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Greater Sudbury, Ontario
  - Research Site, London, Ontario
  - Research Site, North Bay, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- France (4):
  - Research Site, Nice
  - Research Site, Pessac
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Toulouse
- Germany (13):
  - Research Site, Berlin
  - Research Site, Blankenfelde
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Buchholz
  - Research Site, Dülmen
  - Research Site, Frankfurt am Main
  - Research Site, Friedrichshafen
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Kiel
  - Research Site, Münster
  - Research Site, OsnabrÃ¼ck
- Poland (8):
  - Research Site, Iwonicz-Zdrój
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Switzerland (5):
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Zurich

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gottlieb A, Lebwohl M, Liu C, Israel RJ, Jacobson A. Malignancy Rates in Brodalumab Clinical Studies for Psoriasis. Am J Clin Dermatol. 2020 Jun;21(3):421-430. doi: 10.1007/s40257-020-00512-4. PMID 32207067
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total number should be calculated from the induction phase at 661 subjects starting the study. At week 12 if subjects achieved sPGA success (clear[0] or almost clear[1]) they were not continued in the study withdrawal phase to receive drug. Those not achieving success were re-randomized for treatment continuation.
Groups:
- Induction Phase: 210 mg Brodalumab: Administered by subcutaneous (SC) injection until week 12. 210 mg brodalumab: 210 mg brodalumab administered subcutaneous (SC)
- Induction Phase: 140 mg Brodalumab: Administered by subcutaneous (SC) injection until week 12. 140 mg brodalumab: 140 mg brodalumab administered subcutaneous (SC)
- Induction Phase: Placebo: Administered by SC injection until week 12. placebo: Placebo administered subcutaneous (SC)
- Withdrawal Phase: Placebo (140mg): Administered SC injection Week 12 - Week 52
- Withdrawal Phase: 140mg Brodalumab Q2W: Administered SC injection, Week 12 - Week 52
- Withdrawal Phase: Placebo (210mg): Administered SC, Week 12 - Week 52
- Withdrawl Phase: 210mg Brodalumab Q2W: Administered SC injection, Week 12- Week 16
Period: Induction Phase
Arm/Group | Induction Phase: 210 mg Brodalumab | Induction Phase: 140 mg Brodalumab | Induction Phase: Placebo | Withdrawal Phase: Placebo (140mg) | Withdrawal Phase: 140mg Brodalumab Q2W | Withdrawal Phase: Placebo (210mg) | Withdrawl Phase: 210mg Brodalumab Q2W
Started | 222 | 219 | 220 | 0 | 0 | 0 | 0
Completed | 212 | 212 | 209 | 0 | 0 | 0 | 0
Not Completed | 10 | 7 | 11 | 0 | 0 | 0 | 0
Period: Withdrawal Phase
Arm/Group | Induction Phase: 210 mg Brodalumab | Induction Phase: 140 mg Brodalumab | Induction Phase: Placebo | Withdrawal Phase: Placebo (140mg) | Withdrawal Phase: 140mg Brodalumab Q2W | Withdrawal Phase: Placebo (210mg) | Withdrawl Phase: 210mg Brodalumab Q2W
Started (A subset of 283 subjects were rerandomized to Placebo or Brodalumab in the Withdrawal Phase.) | 0 | 0 | 0 | 59 | 57 | 84 | 83
Completed | 0 | 0 | 0 | 6 | 45 | 2 | 74
Not Completed | 0 | 0 | 0 | 53 | 12 | 82 | 9

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Administered by SC injection until week 12. At week 12 participants are assigned to 210 mg brodalumab.
  210 mg brodalumab: 210 mg brodalumab administered subcutaneous (SC)
  placebo: Placebo administered subcutaneous (SC)
- Total: Total of all reporting groups
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo | Total
Number analyzed (Participants) | 222 | 219 | 220 | 661
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (12.2) | 45.8 (13.4) | 46.9 (13.2) | 46.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 57 | 59 | 177
  Male | 161 | 162 | 161 | 484
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 10 | 10 | 8 | 28
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 2 | 5
  Black or African American | 3 | 8 | 6 | 17
  White | 203 | 196 | 202 | 601
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Psoriasis Area and Severity Index (PASI) 75 at Week 12
Description: to evaluate the efficacy of brodalumab (210mg Q2W, 140mg Q2W) in subjects with moderate to severe plaque psoriasis, as measured by the proportion of subjects who achieved 75% improvement in Psoriasis Area Severity Index (PASI75) at week 12.
Time Frame: 0-12 weeks
Population: Data collected is based off of the data from the induction phase.
Measure: Count of Participants; unit: Participants
Groups:
- Induction Phase: 210 mg Brodalumab: Administered by subcutaneous (SC) injection until week 12. At week 12, participants are rerandomized to placebo or continued treatment. Participants are retreated at return of disease.
  210 mg brodalumab: 210 mg brodalumab administered subcutaneous (SC)
  placebo: Placebo administered subcutaneous (SC)
- Induction Phase: 140 mg Brodalumab: Administered by subcutaneous (SC) injection until week 12. At week 12, participants are rerandomized to placebo or continued treatment. Participants are retreated at return of disease.
  140 mg brodalumab: 140 mg brodalumab administered subcutaneous (SC)
  placebo: Placebo administered subcutaneous (SC)
Arm/Group | Induction Phase: 210 mg Brodalumab | Induction Phase: 140 mg Brodalumab | Induction Phase: Placebo
Number analyzed (Participants) | 222 | 219 | 220
Participants | 185 | 132 | 6

2. Primary Outcome: Percentage of Participants With Static Physician Global Assessment (sPGA) Score Success (Score of 0 or 1) at Week 12
Description: To evaluate the efficacy of brodalumab (210mg Q2W, 140mg Q2W) in subjects with moderate to severe plaque psoriasis , as measured by the proportion of subjects who achieved success (clear [0] or almost clear [1]) on the static physicians global assessment (sPGA) at week 12
Time Frame: 0 - 12 Weeks
Population: Data reported is based off of the data collected from the induction phase
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: 210 mg Brodalumab | Induction Phase: 140 mg Brodalumab | Induction Phase: Placebo
Number analyzed (Participants) | 222 | 219 | 220
Participants | 168 | 118 | 3

3. Secondary Outcome: Percentage of Participants With Static Physicians Global Assessment (sPGA) Score Success (Score of 0 or 1) at Week 52
Description: to evaluate maintenance of effect with continued brodalumab treatment (210mg Q2W, 140mg Q2W) as measured by the proportion of subjects achieving success (clear[0] or almost clear [1]) at week 52.
Time Frame: Week 0 - Week 52
Population: Only subjects with efficacy data available at Week 52 were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Withdrawal Phase: Placebo (140mg) | Withdrawal Phase: 140mg Brodalumab Q2W | Withdrawal Phase: Placebo (210mg) | Withdrawl Phase: 210mg Brodalumab Q2W
Number analyzed (Participants) | 6 | 47 | 2 | 72
Participants | 3 | 40 | 0 | 69

ADVERSE EVENTS:
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo
Serious Adverse Events (participants affected / at risk) | 4/222 | 6/219 | 3/220
Other Adverse Events (participants affected / at risk) | 85/222 | 91/219 | 46/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 210 mg Brodalumab (N=222) | 140 mg Brodalumab (N=219) | Placebo (N=220)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis Acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Volvulus of Small Bowel (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Invertebral Disk Intusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 210 mg Brodalumab (N=222) | 140 mg Brodalumab (N=219) | Placebo (N=220)
Upper Respiratory Tract Infection (Infections and infestations) | 18 (18) | 18 (18) | 14 (14)
Headache (Nervous system disorders) | 11 (11) | 12 (12) | 7 (7)
Arthralgia (Injury, poisoning and procedural complications) | 6 (6) | 10 (10) | 6 (6)
Hypertension (Cardiac disorders) | 2 (2) | 8 (8) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 2 (2)
Rhinitis (Infections and infestations) | 5 (5) | 2 (2) | 2 (2)
Tooth Infection (Infections and infestations) | 1 (1) | 6 (6) | 2 (2)
Diarrhoea (Infections and infestations) | 4 (4) | 4 (4) | 1 (1)
Cough (General disorders) | 3 (3) | 6 (6) | 0 (0)
Vomiting (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
Conjunctivitis (Infections and infestations) | 5 (5) | 2 (2) | 0 (0)
Influenza (Immune system disorders) | 4 (4) | 1 (1) | 1 (1)
Myalgia (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Influenza like illness (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Rash (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
UTI (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Dizziness (General disorders) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other